CLINICAL TRIAL: NCT06091995
Title: Use of Belatacept to Delay Tacrolimus Initiation in Kidney Transplant Patients with Delayed Graft Function
Status: Active, not recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 030.PHA.2022.D
Record Dates: First submitted 2023-07-06; First posted 2023-10-23 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Use of Belatacept in Kidney Transplant Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: impact of administering one dose of belatacept on Estimated Glomerular Filtration Rate(eGFR) — Evaluate the clinical impact of administering one dose of belatacept on eGFR at one-year post-transplant, patient and graft survival outcomes, graft rejection, and incidences of BK virus, EBV and CMV infections.
  Other Names: impact of administering one dose of belatacept on eGFR

SUMMARY:
Evaluate the impact of one dose of belatacept in patients with Delayed Graft Function(DGF) on their time to renal recovery and corresponding rates of patient and graft survival, rejection, and incidence of BK virus(BKV), Epstein-Barr Virus(EBV) and/or cytomegalovirus (CMV) infections.

DETAILED DESCRIPTION:
Evaluate the impact of one dose of belatacept in patients with DGF on their time to renal recovery and corresponding rates of patient and graft survival, rejection, and incidence of BK virus, EBV and/or cytomegalovirus (CMV) infections.

At Methodist Dallas Medical Center(MDMC), while providers may choose to initiate belatacept to delay tacrolimus initiation, the impact of this practice on time to renal recovery has not been evaluated. The purpose of this study is to determine if administering belatacept to delay initiation of tacrolimus shortens time to renal recovery in DGF patients

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Received living or deceased donor kidney transplant during study period
* Documented DGF

Exclusion Criteria:

* Multiple organ transplant
* Recipients with acute rejection present on first biopsy evaluation before first belatacept dose
* Recipients with a first dose of belatacept after index discharge or tacrolimus initiation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age ≥18 years Received living or deceased donor kidney transplant during study period Treatment group: kidney transplant recipients with DGF that received belatacept Control group: kidney transplant recipients with DGF that did not receive belatacept
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2025-08-22 (Estimated); Study Completion 2025-08-22 (Estimated)

PRIMARY OUTCOMES:
Time to renal recovery | 1 year
  weeks 1-4, and months 3, 6, 9 and 12) to capture potential short- and long-term effects on renal function.
post-transplant outcome | 1 year
  Patient survival
  o Graft survival Graft rejection

CONTACTS AND LOCATIONS:
Overall Officials: Erin Loncharic, PharmD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI is committed to disseminate research results in a timely fashion. Sharing of data generated by this project will be carried out through presentation at national scientific meetings and/or publication in open access journals. The PI will also make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 2 years
Access Criteria: Clinical trials

REFERENCES:
- [Background] 1. Nulojix (belatacept) [package insert]. Princeton, New Jersey: Bristol-Myers Squibb Company; 2014.
- [Background] Vincenti F, Charpentier B, Vanrenterghem Y, Rostaing L, Bresnahan B, Darji P, Massari P, Mondragon-Ramirez GA, Agarwal M, Di Russo G, Lin CS, Garg P, Larsen CP. A phase III study of belatacept-based immunosuppression regimens versus cyclosporine in renal transplant recipients (BENEFIT study). Am J Transplant. 2010 Mar;10(3):535-46. doi: 10.1111/j.1600-6143.2009.03005.x. PMID 20415897
- [Background] Durrbach A, Pestana JM, Pearson T, Vincenti F, Garcia VD, Campistol J, Rial Mdel C, Florman S, Block A, Di Russo G, Xing J, Garg P, Grinyo J. A phase III study of belatacept versus cyclosporine in kidney transplants from extended criteria donors (BENEFIT-EXT study). Am J Transplant. 2010 Mar;10(3):547-57. doi: 10.1111/j.1600-6143.2010.03016.x. PMID 20415898
- [Background] Jorgenson MR, Descourouez JL, Brady BL, Bowman L, Hammad S, Kaiser TE, Laub MR, Melaragno JI, Park JM, Chandran MM. Alternatives to immediate release tacrolimus in solid organ transplant recipients: When the gold standard is in short supply. Clin Transplant. 2020 Jul;34(7):e13903. doi: 10.1111/ctr.13903. Epub 2020 May 29. PMID 32400907
- [Background] de Graav GN, Baan CC, Clahsen-van Groningen MC, Kraaijeveld R, Dieterich M, Verschoor W, von der Thusen JH, Roelen DL, Cadogan M, van de Wetering J, van Rosmalen J, Weimar W, Hesselink DA. A Randomized Controlled Clinical Trial Comparing Belatacept With Tacrolimus After De Novo Kidney Transplantation. Transplantation. 2017 Oct;101(10):2571-2581. doi: 10.1097/TP.0000000000001755. PMID 28403127